CLINICAL TRIAL: NCT02153216
Title: Formative Phase of Reducing Hazardous Alcohol Use & HIV Viral Load: An RCT in ART Clinics in Vietnam
Brief Title: Formative Phase of Reducing Hazardous Alcohol Use & HIV Viral Load
Acronym: F-REDART
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-0225a; 1R01DA037440-01 (NIH)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Alcohol Drinking; Alcohol Use Norms; Alcohol Use Among ART Clients
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is the Formative Phase of a larger study; once this phase is completed, enrollment into the randomized controlled trial (RCT Phase) will begin. The primary objective of the Formative Phase is to gain a better understanding of the context in which drinking alcohol among ART client in Vietnam occurs, in order to culturally tailor the intervention to be tested in the RCT Phase. Formative Phase activities will consist of up to 40 in-depth interviews with hazardous drinkers who are either: a) ART clients in one of the ART clinics in Thai Nguyen, or b) who are people who inject drugs (PWID) that are not recruited from the ART clinics (whom we will refer to as general population PWID).

ELIGIBILITY:
Inclusion Criteria:

* being 18-49 years of age;
* having an AUDIT score ≥ 8 (hazardous alcohol use);
* being a current ART client at one of the Thai Nguyen ART clinics or a general population PWID;
* being capable of providing voluntary informed consent.

Exclusion Criteria:

* being unable to participate in study activities due to psychological disturbance, cognitive impairment or threatening behavior;
* currently participating in other HIV, drug use or alcohol studies.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ART clients with hazardous alcohol use; PWID in general population with hazardous alcohol use
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Frequency of heavy drinking episodes | during interviews
  This will be an assessment of how and why individuals engage in heavy drinking. As part of this exploration, we will assess:
  * number of standard drinks consumed on those days that an individual drank
  * number of days on which alcohol was consumed beyond recommended levels

CONTACTS AND LOCATIONS:
Overall Officials: Vivian F Go, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Thai Nguyen Center for Preventive Medicine, Thái Nguyên, Thai Nguyen, Vietnam

IPD SHARING:
Plan to Share IPD: No